CLINICAL TRIAL: NCT06302465
Title: Comparison of Narlumosbartmab Combined With Neoadjuvant Chemotherapy and Neoadjuvant Chemotherapy Alone in Bone-derived Malignancies With Osteolytic Lesions and Multinucleated Giant Cells in Local Recurrence Rates: a Prospective, Randomized, Controlled, Two-arm, Open, Single-center Clinical Trial
Brief Title: Narlumosbartmab Combined With Neoadjuvant Chemotherapy in Bone-derived Malignancies With Osteolytic Lesions and Multinucleated Giant Cells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xie Lu, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 18
Record Dates: First submitted 2024-02-25; First posted 2024-03-08 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Malignant Bone Tumor
Keywords: Narlumosbartmab; Malignant bone tumor; Multinucleated giant cell; Osteoclast-like giant cell; Osteolytic; RANKL inhibitor
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant chemotherapy (Active Comparator)
  Interventions: Drug: doxorubicin、cisplatin、methotrexate、ifosfamide
- narlumosbartmab plus neoadjuvant chemotherapy (Experimental)
  Interventions: Drug: narlumosbartmab plus doxorubicin、cisplatin、methotrexate、ifosfamide

INTERVENTIONS:
Drug: narlumosbartmab plus doxorubicin、cisplatin、methotrexate、ifosfamide — Narlumosbartmab is combined with neoadjuvant chemotherapy at 120mg i.h. in day 1, 8, 15, 28 and every 28 days after that.
  Arms: narlumosbartmab plus neoadjuvant chemotherapy
Drug: doxorubicin、cisplatin、methotrexate、ifosfamide — doxorubicin(37.5mg/m^2/d)、cisplatin(120mg/m^2/d)、methotrexate(8-12g/m^2/d)、ifosfamide(2.4g/m^2/d)
  Arms: neoadjuvant chemotherapy

SUMMARY:
Malignant tumor of bone is rare with poor prognosis. Surgery is the main treatment for non- metastatic bone tumor. Although neoadjuvant chemotherapy for non-metastatic bone tumor cannot improve survival rate based on adjuvant chemotherapy, it can reduce and clarify tumor boundary. Control of local recurrence rate is the core objective of oncotherapy. Surgery way and boundary have a significant effect on prognosis of non- metastatic bone tumor. Narlumosbartmab, a RANKL inhibitor, can make tumor boundary clear and reduce surgical difficulty by inhibiting osteoclast. This is a prospective, randomized, controlled, two-arm, open, single-center clinical trial to compare the efficacy and safety of narlumosbartmab combined with neoadjuvant chemotherapy and neoadjuvant chemotherapy alone in bone-derived malignancies with bone lytic lesions and multinucleated giant cells. Investigators mainly observe the local recurrence rate to evaluate the survival benefit for patients with poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age is more than 8 years old and no gender limitation.
2. Histopathologically confirmed high-grade bone-origin malignancies of the limb with the following subtypes: high-grade osteosarcoma, Ewing sarcoma or Ewing sarcoma, malignant giant cell tumor, and undifferentiated pleomorphic sarcoma of bone (the pathological descriptions of the above disease types must include multinuclear giant cell components). Local tumors and isolated lung lesions must be confirmed by pathological diagnosis and multiple lung metastases must be determined by an experienced thoracic surgeon to be resectable.
3. For newly treated tumors that have not been treated with standard therapy and surgery is performed at our center and the necrosis rate is measured.
4. The ECOG physical status score is 0-1, and the expected survival period is more than 6 months.
5. Hb≥ 120g/L，ANC≥1.5×109/L，PLT≥ 100×109/L Cr≤ 1.5×ULN，BUN≤ 2.5×ULN, TB≤ 1.5×ULN, AST and ALT≤ 2.5×ULN, ALB≥ 30 g/L INR）≤1.5，PT and APTT≤1.5×ULN
6. Pregnancy test (urine beta-HCG) negative (for sexually active women of childbearing age).
7. Sign an informed consent form (or legal representative sign) to demonstrate that patients understand the purpose of the study and the procedures required by the study and are willing to participate in the study.

Exclusion Criteria:

1. Past or current jaw osteomyelitis or jaw necrosis; Failure to recover from dental or oral surgery; Acute dental or jaw diseases requiring oral surgery; Those who planned to undergo invasive dental surgery during the study period.
2. Any planned intravenous or oral bisphosphonate therapy during the study period.
3. Past or current use of anti-nuclear factor κB activator ligand (RANKL) antibodies, such as disumab.
4. Metastatic lesions determined by doctors to be unresectable.
5. Have had other malignancies in the past 3 years, are currently being treated with other anti-tumor drugs, or are currently receiving other specific treatments for giant cell tumors of bone (such as radiation, chemotherapy, or embolization).
6. Central nervous system metastases with obvious symptoms, such as headache, brain edema, blurred vision, etc.
7. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite best medical treatment).
8. Patients with grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥450 ms for men and ≥470 ms for women).
9. Patients with grade Ⅲ to Ⅳ cardiac insufficiency according to NYHA criteria, or with left ventricular ejection fraction (LVEF) < 50% indicated by heart color ultrasound, or had myocardial infarction within 6 months before enrollment, or with grade II or above heart failure according to NYHA criteria, uncontrolled angina, uncontrolled severe ventricular arrhythmia, and clinically significant pericardial disease, or electrocardiogram indicates acute ischemia or abnormal active conduction system.
10. Uncontrolled co-morbidities include, but are not limited to poorly controlled diabetes, persistent active infections, or mental illness or social conditions that may affect participants' compliance with the study.
11. Abnormal coagulation function (INR >1.5 or prothrombin time (PT) > ULN+4 seconds or APTT >1.5 ULN), have a tendency to bleed or are receiving thrombolytic or anticoagulant therapy.
12. Patients with a history of psychotropic drug abuse and are unable to quit or have mental disorders.
13. With significant factors affecting the absorption of oral drugs, such as inability to swallow, chronic diarrhea and intestinal obstruction.
14. Patients with active viral hepatitis B or hepatitis C, or those with active infections requiring antimicrobial treatment (e.g. antibiotics, antiviral drugs, antifungal drugs).
15. Have participated in clinical trials of other antitumor drugs within 4 weeks.
16. Known allergic reactions, hypersensitivities, or intolerances to chemotherapy agents or their excipients.
17. During lactation.
18. Patients received vaccination during the course of treatment, or within 4 weeks of vaccination.
19. Any condition which, in the opinion of the investigator, is likely to harm the subject or cause the subject to be unable to meet or perform the study requirements.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
local recurrence rate | 2 years

SECONDARY OUTCOMES:
tumor necrosis rate | 12 weeks
R0 removal rate | 12 weeks
  R0 remove mains the pathological margin is negative.
Event-free survival | 2 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lu Xie, M.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China